CLINICAL TRIAL: NCT06264752
Title: Multi-hospital Electronic Decision Support for Drug-associated Acute Kidney Injury (MEnD-AKI)
Brief Title: Multi-hospital Electronic Decision Support for Drug-associated Acute Kidney Injury
Acronym: MEnD-AKI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: University of Florida (Other); University of Pittsburgh Medical Center (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Sandra Kane-Gill, PharmD, MSc, FCCP, FCCM, Professor of Pharmacy, Department of Pharmacy and Therapeutics, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY20120008; R01DK121730 (NIH)
Record Dates: First submitted 2024-02-08; First posted 2024-02-20 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Acute Kidney Injury
Keywords: acute kidney injury; drug-associated acute kidney injury; adverse drug event; pharmacist
MeSH Terms: conditions — Acute Kidney Injury; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, interventional controlled trial at eight hospitals within the UPMC health-system. Researchers will randomize 38 hospital service clusters to receive either: 1) a Cerner electronic medical record (EMR)-based AKI passive alert which is standard of care at UPMC: this alert provides decision support within the EMR for the diagnosis and basic staging of AKI but without specific recommendations for management (Usual Care Arm); or 2) protocolized stage-based intervention delivered to the physician by a pharmacist for consideration and approval. Hospital service clusters will be allocated 1:1 to the intervention or usual care with a web-based system to maintain concealment using a randomized block design.
Who Masked: Outcomes Assessor
Masking Description: Statisticians performing the analysis will be blinded to the treatment allocation.
  The investigators will randomize clusters to intervention and control within strata defined hospitals to adjust for inherent subgroup differences. The allocation sequence list will be maintained by the data management team (DMT) using a secure web-based system where assignments will be maintained and accessed by the CDSS. Pharmacists will only receive alerts for patients of physicians randomized to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Protocolized stage-based intervention (Experimental): The intervention uses an automated alerting system to identify patients: 1) receiving a high-risk drug or drug combination associated with AKI and at low-risk for progression to either stage 2 AKI or stage 3 AKI (Level A) and 2) patients without AKI or stage 1 AKI receiving a high-risk drug or drug combination associated with AKI and at high risk for progression to either stage 2 AKI or stage 3 AKI, and patients with AKI stage 2 or stage 3 receiving a high-risk drug or drug combination associated with AKI or a medication that requires renal dose adjustment (Level B). This patient specific risk-profile will be coupled with recommendations for medication management and delivered to the physician by a pharmacist for consideration and approval.
  Interventions: Other: Level A; Other: Level B
- Usual Care (Active Comparator): A Cerner EMR-based AKI passive alert which is standard of care at UPMC.
  Interventions: Other: Passive Alert

INTERVENTIONS:
Other: Level A — Pharmacy personnel will generate a general recommendation based on the AKI KDIGO management guidelines to the physician.
  Arms: Protocolized stage-based intervention
Other: Level B — The pharmacist will make nephrotoxic/renally eliminated medication management recommendations to the attending physician (or designee). Recommendations may include stopping or changing a drug, changing dose or schedule, ordering laboratory tests, taking no action, or other. The pharmacist will record details of the interaction with the physician and whether recommendations were accepted.
  Arms: Protocolized stage-based intervention
Other: Passive Alert — Passive Cerner alert provides decision support within the EMR for the diagnosis and basic staging of AKI but without specific recommendations for management.
  Arms: Usual Care

SUMMARY:
This study is a randomized controlled trial at eight hospitals within the University of Pittsburgh Medical Center-UPMC system. The project will assess the efficacy of a clinical surveillance system augmented with near real-time predictive analytics to support a pharmacist-led intervention delivered to attending physicians (primary service) to reduce the progression and complications of drug-associated acute kidney injury (D-AKI) in hospitalized (non-ICU) adults.

DETAILED DESCRIPTION:
Researchers will randomize 38 hospital service clusters to receive either: 1) a Cerner electronic medical record (EMR)-based AKI passive alert which is standard of care at UPMC: this alert provides decision support within the EMR for the diagnosis and basic staging of AKI but without specific recommendations for management (Usual Care Arm); or 2) protocolized stage-based intervention delivered to the physician by a pharmacist for consideration and approval. The intervention uses an automated alerting system to identify patients: 1) receiving a high-risk drug or drug combination associated with D-AKI and at low-risk for progression to either stage 2 AKI or stage 3 AKI per KDIGO criteria (Level A) and 2) patients without AKI or stage 1 AKI receiving a high-risk drug or drug combination associated with D-AKI and at high risk for progression to either stage 2 AKI or stage 3 AKI per KDIGO criteria, and patients with AKI stage 2 or stage 3 receiving a high-risk drug or drug combination associated with D-AKI or a medication that requires renal dose adjustment (Level B). This patient specific risk-profile will be coupled with recommendations for medication management and delivered to the physician by a pharmacist for consideration and approval. Additionally, the investigators will assess cost-effectiveness and physicians' perception of the pharmacist-led service.

The primary outcome is Major Adverse Kidney Events within 30 days of randomization (MAKE30), defined as defined as a composite of death, new kidney replacement therapy, or final serum creatinine ≥150% of reference at the earliest of hospital discharge or 30 days from study enrollment, whichever occurs first. Key secondary outcomes include: progression of AKI from time of Level B intervention (first alert generated) to hospital discharge, AKI intensity (duration of AKI by all stages, duration of AKI stage 2, and duration of AKI stage 3), and nephrotoxic burden.

ELIGIBILITY:
Inclusion Criteria:

Physician-subject Inclusion

* Physicians employed at UPMC hospital systems
* Attending physicians of record who care for patients across multiple units outside ICU/ED
* Physician cares for 1 or more patient receiving a system alert identifying high-risk for AKI

Patient-subject Inclusion

* System alert identifying risk for AKI
* Patient has attending physician who is participating in the randomized clusters
* After initial patient inclusion, an individual patient will not be eligible for re-inclusion until after 90 days. Re-inclusion will only be allowed if a separate hospital admission/encounter occurs and only starting on day 91

Exclusion Criteria:

Physician-subject Exclusion

* Physicians of record who only care for ICU or ED patients
* Physicians who primarily provide care for transplant (heart, kidney, liver, etc.) patients
* Physicians who primarily provide consult services only (dermatology, rehabilitation, etc.)

Patient-subject Exclusion

• Patients with end stage renal disease on admission, baseline eGFR <15, comfort measures only, or died before the intervention could be delivered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 698 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Major Adverse Kidney Events within 30 days of randomization (MAKE30) | up to 30 days
  Composite of death, new kidney replacement therapy, or final serum creatinine greater than or equal to 150 percent of reference at the earliest of hospital discharge or 30 days from study enrollment, whichever occurs first.

SECONDARY OUTCOMES:
Progression of AKI from time of Level B intervention (first alert generated) to hospital discharge | up to 30 days
  Percentage of high-risk patients without AKI at the time of a first level B alert who subsequently progress to maximum AKI severity stages 1, 2, or 3 before hospital discharge or 30 days, whichever comes first.
  Percentage of high-risk patients diagnosed with stage-1 AKI at the time of a level B alert who subsequently progress to maximum severity stages 2 or 3 AKI before hospital discharge or 30 days, whichever comes first.
  Percentage of high-risk patients diagnosed with stage-2 AKI at the time of a level B alert who subsequently progress to maximum severity stage 3 AKI before hospital discharge or 30 days, whichever comes first.
AKI Intensity: Duration of AKI for all stages; Duration of AKI Stage 2; Duration of AKI stage 3 | up to 30 days
  AKI intensity rate (per 100 exposed patient-days) calculated as:
  number of days patients have AKI/ total number of AKI exposed patient-days standardized per 100 exposed days
Nephrotoxic burden | up to 30 days
  Drug.days* in both study arms for those drugs considered possible/probable, probable and definitely related to AKI in adult, non-ICU patients.
  *Drug.days calculation: each drug and each day of therapy increases the burden by 1 drug.day.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra L Kane-Gill, PharmD, MS, Principal Investigator — University of Pittsburgh; Azra Bihorac, MD, MS, Principal Investigator — University of Florida
Locations (8):
- United States (8):
  - UPMC Altoona, Altoona, Pennsylvania
  - UPMC Horizon, Farrell, Pennsylvania
  - UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC Jameson, New Castle, Pennsylvania
  - UPMC Magee, Pittsburgh, Pennsylvania
  - UPMC Presbyterian/Montefiore, Pittsburgh, Pennsylvania
  - UPMC Shadyside, Pittsburgh, Pennsylvania
  - UPMC Williamsport, Williamsport, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stottlemyer BA, Kellum JA, Bihorac A, Ozrazgat-Baslanti T, Murugan R, Chang CH, Amatullah N, Tran TL, Lukan CJ, Elder MM, Adiyeke E, Ren Y, Ricketts D, Emanuele B, Rashidi P, Kane-Gill SL. Multi-hospital electronic decision support for drug-associated acute kidney injury (MEnD-AKI): Study protocol for a randomized clinical trial. Contemp Clin Trials. 2025 Oct;157:108055. doi: 10.1016/j.cct.2025.108055. Epub 2025 Aug 22. PMID 40850370